CLINICAL TRIAL: NCT04580212
Title: Improving Hygienic Management of Poultry in Rural Uganda
Brief Title: Poultry Management and Child Diarrhea in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: The Water Trust (Unknown)
Responsible Party: Principal Investigator, Ayse Ercumen, Assistant Professor, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 698
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators and data analysts will be blinded to intervention assignment by using a numerical code for study arm during analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): This arm received the poultry hygiene intervention.
  Interventions: Behavioral: Poultry hygiene intervention
- Control arm (No Intervention): This arm received no intervention.

INTERVENTIONS:
Behavioral: Poultry hygiene intervention — The intervention will consist of a series of participatory training exercises designed to accomplish three main goals: (1) increase awareness of health risks and lost livelihood benefits of current poultry management practices, (2) build practical skills for poultry management, and (3) build supportive community norms by facilitating savings group discussions on poultry management. The intervention will be delivered through three activities: (1) triggering exercise designed to raise awareness of both the health risks of the current practices and the economic potential of a more active poultry management approach, and ultimately to motivate participants for behavior change, (2) poultry management training activity based on local needs and norms, and (3) periodic follow-on coaching to reinforce messages from the initial training and emphasize action planning, monitoring of plan execution, and troubleshooting.
  Arms: Intervention arm

SUMMARY:
Fecal contamination from animal sources, specifically chickens, is increasingly recognized as a risk factor for enteric infections in low-income countries where domestic animals are often kept in close proximity to living quarters. Community members typically allow chickens to move freely around their compound and in their homes. Unlike other animals, such as cows or goats, poultry are typically not confined and their feces, which are relatively small, are considered relatively innocuous and therefore largely ignored by adults and children. In this study, the investigators have implemented an intervention to help rural poultry owners with children to hygienically separate chickens from children by focusing on a small set of key factors, including increased risk perception, increased perception of potential livelihood benefits, increased skills, and increased supportive social norms. The investigators hypothesized that the poultry hygiene intervention will lead to improved poultry management practices, which will in turn lead to reduced fecal contamination in the domestic environment and subsequently reduced diarrheal illness in young children. To measure these parameters along the causal chain, the investigators used a combination of household surveys, spot check observations and testing of environmental samples for fecal contamination.

ELIGIBILITY:
Inclusion Criteria:

* At least one person in the household is a member of Self-Help Groups formed by The Water Trust, Uganda
* There is at least one child under the age of 5 years living in the household
* There is an adult (>18 years) primary caregiver of a child <5 years available for participation in study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of children <5 years with caregiver-reported diarrhea in past 7 days | Caregiver reported 7-day prevalence of diarrhea in children <5 years, measured approximately 1 year after initiation of intervention
  Diarrhea defined as 3 or more soft or watery stools in 24-hour period

SECONDARY OUTCOMES:
Proportion of households with E.coli in household environmental samples | Ascertained with analysis of samples from households, collected approximately 1 year after initiation of intervention
  Detection of E. coli (general fecal indicator)
Proportion of households with observed poultry feces in compound | Ascertained by spot check observation approximately 1 year after initiation of intervention
  Poultry feces occurrences observed in household compounds

OTHER OUTCOMES:
Prevalence of children <5 years with caregiver-reported respiratory infection in past 7 days | Caregiver reported 7-day prevalence of respiratory infection in children <5 years, measured approximately 1 year after initiation of intervention
  Respiratory infection defined as any of the following symptoms: Constant cough, congestion, runny nose, panting, wheezing, or difficulty breathing

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ercumen, Principal Investigator — North Carolina State University; Angela Harris, Principal Investigator — North Carolina State University; Chris Prottas, Study Director — The Water Trust
Locations (1):
- The Water Trust, Kampala, Uganda